CLINICAL TRIAL: NCT02431845
Title: Pharmaco(Epi)Genetic, Proteomic, and Microbiomic Study of Obsessive-Compulsive
Brief Title: Pharmaco(Epi)Genetic, Proteomic, and Microbiomic Study of Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Se Joo Kim, Professor, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0577 and 4-2015-0655
Record Dates: First submitted 2015-04-23; First posted 2015-05-01 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Pharmaco(epi)genetics; Microbiome; Proteome
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Intervention Model Description: Open naturalistic treatment
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SSRIs treatment as usual OCD gruop (Experimental): SSRIs treatment as usual fluoxetine 40~80 mg dose equivalent (fluoxetine, paroxetine, sertraline, fluvoxamine, escitalopram, clomipramine)
  Interventions: Drug: SSRIs

INTERVENTIONS:
Drug: SSRIs — usual dose SSRI for obsessive-compulsive disorder, i.e. fluoxetine 40~80 mg dose equivalents
  Other Names: five kinds of SSRIs including fluoxetine

SUMMARY:
The purpose of this study is to determine whether pharmaco(epi)genetic study predict selective serotonin reuptake inhibitor (SSRI) responsiveness in advance before the appearance of the drug effect until 4 months(16 weeks), 6 months, and 1 year after administration of SSRIs.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of (epi)genetic variants on the response to SSRIs in obsessive-compulsive disorder (OCD) subject.

The investigators will recruit drug-naive or drug-free(> 3 months) OCD subjects (n=200). The participants will get SSRIs for their OCD symptoms. The type and dose of SSRIs will not be restricted and will depend on the individual participant's state. However, the investigators will be recommended to follow usual clinical guideline (the Korean treatment algorithm for OCD, 2004). At baseline, 4 month, 6 months, and 1 year after treatment, the participants will be evaluated by Yale-Brown Obsessive-Compulsive Scale(YBOCS), Montgomery Asberg Depression Rating Scale(MADRS), Dimensional Obsessive-Compulsive Scale(DOCS), Toronto alexithymia scale (TAS), interpersonal reactivity index (IRI), Barratt impulsiveness scale (BIS), and the Measure of Constructs Underlying Perfectionism(M-CUP), Beck Depression Inventory(BDI), Beck Anxiety Inventory(BAI), Intolerance of Uncertainty (IOU), Metacognition, Disgust scale, Early Trauma Inventory (ETI). And a part of participants will be taken resting state functional MRI.

The research participants will donate approximately 10-15 ml of blood, from which we will extract DNA and separate serum. Using various (epi)genetic analyses, proteomics, and microbiome analysis (circulating bacterial extracellular vesicles) methods, we will analyze the association of various (epi)genetic variants, protein profiles, microbiome and the anti-obsessive-compulsive responses.

ELIGIBILITY:
Inclusion Criteria:

1. age 19~ 70
2. OCD by Diagnostic and Statistical Manual for Mental disorders, 4th edition (DSM-IV)
3. drug naive or drug free for more than 3 months

Exclusion Criteria:

1. any neurological disorder
2. comorbid psychotic disorders
3. alcohol or other substance dependence within past 6 months
4. any evidences for brain diseases

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Yale-Brown Obsessive-Compulsive Scale | baseline, 3 or 4 months, 6 months, 1 year
  rating scale for obsessive-compulsive symptom severity consisting of 10 items

SECONDARY OUTCOMES:
Change from the baseline Montgomery-Asberg Depression Rating Scale | baseline, 3 or 4 months, 6 months, 1 year
  rating scale for depressive symptom severity consisting of 10 items, Various psychometric characteristics
Occurrence of any side effects during the SSRIs treatment | 3 or 4 months, 6 months, 1 year
  any adverse events related to SSRI use

CONTACTS AND LOCATIONS:
Overall Officials: Se Joo Kim, M.D., Principal Investigator — Professor, Department of Psychiactry, Yonsei Univ. College of Medicine
Locations (1):
- Yonsei Univ. Health System Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No